CLINICAL TRIAL: NCT02710734
Title: A Phase II Trial of Risk Enabled Therapy After Initiating Neoadjuvant Chemotherapy for Bladder Cancer (RETAIN BLADDER)
Brief Title: Risk Enabled Therapy After Initiating Neoadjuvant Chemotherapy for Bladder Cancer (RETAIN)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GU-086; 15-1071 (Other: Fox Chase Cancer Center IRB)
Record Dates: First submitted 2016-02-18; First posted 2016-03-17 (Estimated); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Urothelial Carcinoma of the Bladder
Keywords: Urothelial
MeSH Terms: interventions — Methotrexate; Vinblastine; Doxorubicin; Cisplatin; Radiotherapy, Intensity-Modulated; Transurethral Resection of Bladder; Fluorouracil; Mitomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- CRT (Experimental): Trimodality of Maximal TURBT#1 Followed by AMVAC and TURBT#2 and then chemoradiation followed by TURBT#3
  Interventions: Drug: Methotrexate; Drug: Vinblastine; Drug: Doxorubicin; Drug: Cisplatin; Radiation: Intensity modulated radiation therapy (IMRT); Procedure: Transurethral Resection of Bladder tumor; Drug: 5-FU; Drug: Mitomycin C
- Surveillance (Experimental): Trimodality of Maximal TURBT#1 Followed by AMVAC and TURBT#2 and then active surveillance
  Interventions: Drug: Methotrexate; Drug: Vinblastine; Drug: Doxorubicin; Drug: Cisplatin; Procedure: Transurethral Resection of Bladder tumor
- Intravesicle therapy (Experimental): Trimodality of Maximal TURBT#1 Followed by AMVAC and TURBT#2 and then intravesicle therapy followed by TURBT#3
  Interventions: Drug: Methotrexate; Drug: Vinblastine; Drug: Doxorubicin; Drug: Cisplatin; Procedure: Transurethral Resection of Bladder tumor
- Radical Cystectomy (Experimental): Trimodality of Maximal TURBT#1 Followed by AMVAC and TURBT#2 and then cystectomy
  Interventions: Drug: Methotrexate; Drug: Vinblastine; Drug: Doxorubicin; Drug: Cisplatin; Procedure: Transurethral Resection of Bladder tumor

INTERVENTIONS:
Drug: Methotrexate — Administered Day 1 of each 14 day cycle for 3 cycles
Drug: Vinblastine — Administered Day 1 of each 14 day cycle for 3 cycles
Drug: Doxorubicin — Administered Day 1 of each 14 day cycle for 3 cycles
Drug: Cisplatin — Administered Day 1 of each 14 day cycle for 3 cycles
Radiation: Intensity modulated radiation therapy (IMRT) — 2.0 Gy per fraction to the whole bladder plus a margin for a total of 32 fractions (64.0 Gy). Radiation will be administered from Monday to Friday
  Arms: CRT
Procedure: Transurethral Resection of Bladder tumor — Performed at before and after AMVAC and after chemoradiation and intravesicle therapy
Drug: 5-FU — Continuous 24hr Intravenous infusion days 1-5 and 16-20 with radiation treatment
  Arms: CRT
Drug: Mitomycin C — Intravenous on day 1 with radiation treatment
  Arms: CRT

SUMMARY:
The aim of this study is to evaluate a risk-adapted approach to the treatment of muscle invasive bladder cancer. Each baseline transuretheral resection of bladder tumor (TURBT) sample will be sequenced while proceeding with neoadjuvant accelerated methotrexate, vinblastine, doxorubicin, and cisplatin (AMVAC) chemotherapy. Based on the mutational profile and the post AMVAC TURBT findings, patients will be treated with active surveillance (experimental arm), or standard of care intravesicle therapy, chemoradiation or surgery. We hypothesize that this approach will lead to non-inferior metastasis-free survival at 2 years, while preserving the bladder and thus quality-of-life for a proportion of patients.

DETAILED DESCRIPTION:
This phase II trial studies how well maximal transurethral surgery (surgery performed with a special instrument inserted through the urethra) followed by accelerated methotrexate, vinblastine, doxorubicin hydrochloride, cisplatin, and radiation therapy work in treating patients with bladder cancer that has spread to the muscle. Drugs used in chemotherapy, such as methotrexate, vinblastine sulfate, doxorubicin hydrochloride, and cisplatin work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Radiation therapy uses high-energy x-rays to kill tumor cells and shrink tumors. Giving chemotherapy with radiation therapy may kill more tumor cells. Giving combination chemotherapy and radiation therapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥18 years.
* Primary urothelial or predominantly urothelial carcinoma of the bladder.
* Histologic evidence of muscularis propria invasion.
* AJCC27 clinical stage T2-T4a .
* No radiographic evidence of lymph node positivity (N0) or metastatic disease (M0). Clinical lymphadenopathy on staging CT greater than 1.5 cm in short axis must be biopsy proven negative.
* ECOG performance status 0, 1, or 2.
* Left ventricular ejection fraction ≥ 50% by MUGA or ECHO within 6 months of study entry.
* Normal organ and bone marrow function as defined:

Leukocytes ≥ 3,000/mcL Absolute neutrophil count ≥ 1,500/mcL Platelets ≥ 100,000/mcL Total bilirubin ≤ institutional upper limit of normal (ULN) AST(SGOT)/ALT(SGPT) ≤ 2.5 X institutional ULN Creatinine Creatinine Clearance ≥ 50 mL/min (calculated using the Cockroft-Gault formula or measured with 24 hour urine collection)

Exclusion Criteria:

* Any component of small cell histology.
* Prior pelvic radiation therapy or patients who have undergone prior radiation to greater than or equal to 25% of the bone marrow within the past year are excluded due to risk of life threatening myelosuppression
* Prior systemic chemotherapy; patients who have received any previous systemic chemotherapy or radiation therapy for urothelial carcinoma or cytotoxic chemotherapy for another malignancy within 1 year of study entry are ineligible.
* Prior or concurrent malignancy of any other site except for non-melanoma skin cancer, unless disease free interval ≥ 5 years.
* Patients who have received experimental agents within 4 weeks of study entry.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Methotrexate, Vinblastine, Adriamycin or Cisplatin or other agents used in the study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection (defined by current oral or intravenous antibiotic therapy), symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study due to the potential for teratogenic or abortifacient effects of cytotoxic chemotherapy.
* Known HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with cytotoxic chemotherapy. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy.
* Patients with hydronephrosis that has not been addressed with an intervention such as placement of a stent.
* Pregnancy & Women of Childbearing Potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2016-02-24 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2034-02 (Estimated)

PRIMARY OUTCOMES:
Metastasis-free survival (MFS) at 2 years. | 24 months

SECONDARY OUTCOMES:
Ability to complete of 3 cycles of neoadjuvant AMVAC and chemoradiation therapy with 5-FU and mitomycin C. | Up to 37 Weeks

OTHER OUTCOMES:
Rate of urothelial carcinoma recurrence in active surveillance patients | 60 months
Overall survival and PFS of the entire cohort | 60 months
toxicity during each treatment arm according to NCI CTCAE v 4.01 criteria | 24 months
Proportion of patients with ≥cT1 disease after TURBT#2 | up to 22 weeks
Proportion of patients requiring a cystectomy, either immediately after TURBT#2 or as salvage after surveillance or CRT | up to 24 months
Endoscopic Tumor Quantification System score at each TURBT | 24 months
  At each cystoscopic examination, the location and extent of tumor volume will be visually depicted and graded according to Endoscopic Tumor Quantification System
Quality of life with neoadjuvant AMVAC and subsequent risk-adapted treatment | 60 months
  American Urologic Association (AUA) Symptom Index Score, Sexual Health Inventory for Men (SHIM) score or Female Sexual Function Index (FSFI) score

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Washington Cancer Institute at MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Johns Hopkins, Baltimore, Maryland
  - Sidney kimmel Cancer Center, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Geynisman DM, Abbosh PH, Ross E, Zibelman MR, Ghatalia P, Anari F, Mark JR, Stamatakis L, Hoffman-Censits JH, Viterbo R, Greenberg RE, Churilla TM, Horwitz EM, Hallman MA, Smaldone MC, Uzzo R, Chen DYT, Kutikov A, Plimack ER. Phase II Trial of Risk-Enabled Therapy After Neoadjuvant Chemotherapy for Muscle-Invasive Bladder Cancer (RETAIN 1). J Clin Oncol. 2025 Mar 20;43(9):1113-1122. doi: 10.1200/JCO-24-01214. Epub 2024 Dec 16. PMID 39680823
- [Derived] Jiang DM, Chung P, Kulkarni GS, James ND, Sridhar SS. Lack of Evidence Does Not Equal Lack of Benefit: Neoadjuvant Chemotherapy and Trimodality Therapy in Selected Patients with Muscle-Invasive Bladder Cancer : In response to: Dirk Bohmer and Arne Grun. Lacking Evidence to Recommend Neoadjuvant Chemotherapy and Definitive Radiotherapy in Muscle-Invasive Bladder Cancer. Curr Oncol Rep. 2021 Mar 3;23(3):36. doi: 10.1007/s11912-021-01035-9. No abstract available. PMID 33660142